CLINICAL TRIAL: NCT02487524
Title: Biomarkers of Neuropathic Pain in Women Treated for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: deCODE genetics (Industry)
Responsible Party: Principal Investigator, Hanna Harno, MD, PhD, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 149/13/03/00/14
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Neuropathic Pain; Breast Cancer
Keywords: Neuropathic Pain; Breast Cancer; Post surgical
MeSH Terms: conditions — Neuralgia; Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nerve resection with pain (Other): Questionnaires, cognitive tests, sensory examination, cold water test with autonomic nervous system monitoring. QST.
  Interventions: Other: Cold water test; Other: Autonomic nervous system monitoring; Other: QST
- Nerve resection without pain (Other): Questionnaires, cognitive tests, sensory examination, cold water test with autonomic nervous system monitoring. QST.
  Interventions: Other: Cold water test; Other: Autonomic nervous system monitoring; Other: QST
- No nerve resection but pain (Other): Questionnaires, cognitive tests, sensory examination, cold water test with autonomic nervous system monitoring. QST.
  Interventions: Other: Cold water test; Other: Autonomic nervous system monitoring; Other: QST

INTERVENTIONS:
Other: Cold water test — The patients immerse their hand into cold water for a maximum of 90 seconds and report their pain intensity every 15 seconds during the test.
Other: Autonomic nervous system monitoring — The autonomic nervous system is monitored during the cold water test and 15 minutes thereafter.
Other: QST — Quantitative sensory testing.

SUMMARY:
Investigators aim to identify the key phenotypes (biological, psychological, genetic) involved in the transition from acute to chronic neuropathic pain (NP) by comparison of the neuropathic pain phenotypes and genomics of patients developing NP or not under similar nerve injury conditions. The cohort is part of a previous prospective study of 1000 patients operated for breast cancer of whom 350 have surgeon defined intercostobrachial nerve resection during operation with or without persistent pain and additional 50 patients with pain, but no nerve resection during operation. Patients fill in questionnaires and a detailed sensory examination, cognitive tests, and a cold water test with autonomic nervous system monitoring are performed during the research visit. A selected group of patients undergo quantitative sensory testing (QST).

DETAILED DESCRIPTION:
This cohort is part of a previous prospective study of 1000 breast cancer operated women. Of these, there are 350 patients with surgeon defined intercostobrachial nerve resection during the operation. Part of the patients have pain, part of them are pain free. In addition the investigators plan to enroll 50 patients with pain, but no nerve resection during operation.

The patients come for a clinical research visit. Beforehand they fill in questionnaires of medical history, pain, mood, temperament, quality of life, and sleeping. After informed consent the patients give a blood sample with prior 12 hour fasting. The investigators present a detailed sensory testing with body maps and patient pain drawings. The investigators perform a cold water test with autonomic nervous system monitoring and conduct a set of cognitive tests, part of them computer based. A selected group of patients undergo QST.

ELIGIBILITY:
Inclusion Criteria:

* belongs to the cohort of 1000 breast cancer operated women and has had nerve resection during the operation (with or without pain) or no nerve resection, but pain
* sufficient Finnish language skills

Exclusion Criteria:

* age over 75 years
* living far away from study site

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

PRIMARY OUTCOMES:
Composite factors related to the persistence of pain after nerve injury | 5 years
  Study of associations between phenotypic and genotypic data. Phenotyping is assessed by detailed sensory testing, questionnaires related to pain (Brief Pain Inventory, Numeric Rating Scale), psychological factors (Pain Catastrophizing Scale, Hospital Anxiety and Depression Rating Scale), personality (Ten-item Personality Inventory) and quality of life (36-item Short Form Health Survey and Insomnia Severity Index). Additionally, cognitive tests, a cold water test with autonomic nervous function monitoring, and a blood sample. DNA will be isolated from blood samples and analyzed for genetic variants associated with new neuropathic pain phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Eija Kalso, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, HUS, Finland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Kaunisto MA, Jokela R, Tallgren M, Kambur O, Tikkanen E, Tasmuth T, Sipila R, Palotie A, Estlander AM, Leidenius M, Ripatti S, Kalso EA. Pain in 1,000 women treated for breast cancer: a prospective study of pain sensitivity and postoperative pain. Anesthesiology. 2013 Dec;119(6):1410-21. doi: 10.1097/ALN.0000000000000012. PMID 24343286
- [Background] Meretoja TJ, Leidenius MHK, Tasmuth T, Sipila R, Kalso E. Pain at 12 months after surgery for breast cancer. JAMA. 2014 Jan 1;311(1):90-92. doi: 10.1001/jama.2013.278795. No abstract available. PMID 24381969
- [Background] Haanpaa M, Attal N, Backonja M, Baron R, Bennett M, Bouhassira D, Cruccu G, Hansson P, Haythornthwaite JA, Iannetti GD, Jensen TS, Kauppila T, Nurmikko TJ, Rice ASC, Rowbotham M, Serra J, Sommer C, Smith BH, Treede RD. NeuPSIG guidelines on neuropathic pain assessment. Pain. 2011 Jan;152(1):14-27. doi: 10.1016/j.pain.2010.07.031. Epub 2010 Sep 19. PMID 20851519
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Derived] Aho T, Sipila R, Kalso E, Harno H. Temperament and character dimensions differ in chronic post-surgical neuropathic pain and cold pressure pain. Scand J Pain. 2022 Feb 9;22(3):515-525. doi: 10.1515/sjpain-2021-0163. Print 2022 Jul 26. PMID 35139264
- [Derived] Honkanen N, Mustonen L, Kalso E, Meretoja T, Harno H. Breast reconstruction after breast cancer surgery - persistent pain and quality of life 1-8 years after breast reconstruction. Scand J Pain. 2021 Jun 7;21(3):522-529. doi: 10.1515/sjpain-2021-0026. Print 2021 Jul 27. PMID 34087967
- [Derived] Sipila R, Kemp H, Harno H, Rice ASC, Kalso E. Health-related quality of life and pain interference in two patient cohorts with neuropathic pain: breast cancer survivors and HIV patients. Scand J Pain. 2021 Mar 17;21(3):512-521. doi: 10.1515/sjpain-2020-0177. Print 2021 Jul 27. PMID 33725747